CLINICAL TRIAL: NCT04720508
Title: Aberrant Expression of Circulating Micro RNA as a Biomarker for Diagnosis of Breast Cancer in Egyptian Females
Brief Title: Aberrant Expression of Micro RNA for Diagnosis of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hosam Atif Sayed Anas, Principal Investigator, Assiut University
Other Study IDs: miRNA in breast cancer
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (patient group): included 25 patients with BC admitted to department of medical Oncology, South Egypt Cancer Institute, Assiut University.
  blood samples will be obtained after getting informed consent.
  Interventions: Diagnostic Test: blood sample collection.
- Group B (control group): included 25 controls age-matched , sex-matched and apparently healthy. blood samples will be obtained after getting informed consent .
  Interventions: Diagnostic Test: blood sample collection.

INTERVENTIONS:
Diagnostic Test: blood sample collection. — venipuncture procedure

SUMMARY:
In this study we aim to:

1. Assess serum miRNA-373, miRNA-425-5p expression in patients with breast cancer.
2. Explore their correlations with breast cancer clinicopathological documented data including staging, grading and tumor receptors.

DETAILED DESCRIPTION:
Breast cancer (BC) is the leading cause of cancer worldwide with estimated 2.3 million new cases and 685000 deaths in 2020. In women, breast cancer accounts for one in 4 cancer cases and one in 6 cancer deaths.

In Egypt, BC is the most common cancer among females accounting for 32.0% of all cancers in women according to the data of the National Cancer Registry Program of Egypt . 22038 Egyptian females breast cancer new cases were estimated to be in 2020 .

The most important risk factors for breast cancer include female gender, age (30 years old and older), positive family history for breast cancer , and familial genetic mutations, including mutations in the breast cancer A1 (BRCA1) and BRCA2 genes. Furthermore, women with a history of breast cancer are more likely (20-25%) to develop microscopic cancer in the opposite breast. A positive history for cancer in the endometrium, ovaries, or colon, as well as radiation therapy for Hodgkin's lymphoma, was shown to increase the risk of breast cancer.

The gold standard for diagnosis of breast cancer is histopathology. Several tumor markers have been suggested for the evaluation and management of breast cancer including estrogen and progesterone receptors (ER/PR), which are used for the assessment of susceptibility to hormone treatment, and human epidermal growth factor receptor 2 (HER2), which is used to assess the susceptibility to trastuzumab treatment.

With the rapid development of medical technology, strategies such as surgery, medication and radiotherapy can help a lot to reduce mortality rate. Though clinical intervention at early stage can greatly improve prognosis, many BC patients are asymptomatic until disease progression.

Thus, effective screening methods are in great demand for the early detection of BC. In clinical practice, many screening strategies have been widely used, such as mammography, breast magnetic resonance imaging (MRI) and ultrasound imaging.

However, these strategies are far from being perfect because of over-diagnosis, false-positive inconsistent results and potential radiation injury.

Core needle aspiration can help establish the diagnosis, but the procedure is invasive and not suitable for routine use .

Therefore, novel non-invasive screening methods of high sensitivity and specificity are needed to assist the early diagnosis of BC .

Microribonucleic Acids (microRNAs) are a large subgroup of noncoding RNAs made up of 18-25 nucleotides. MicroRNAs regulate gene expression after transcription. They have a multifunctional role, as they can perform either as oncogenes by repressing their target tumor suppressor genes, or as tumor suppressors through inhibiting the expression of their target oncogenes.

Numerous studies have shown that miRNAs played important roles in nearly all biological processes and their aberrant expression was associated with many diseases including cancers. Stable existence of miRNAs in peripheral blood circulation revealed that they could be promising noninvasive biomarkers for cancer detection.

For BC, more and more circulating miRNAs (ie, miRNA-373, miRNA-425-5p) are emerging as potential diagnostic or prognostic biomarkers.

In breast cancer miRNA-425-5p was found elevated and predicted a poor prognosis for the patients, and its role in BC highlight a new research points for diagnostic and therapeutic plans.

MiRNA-373 Circulating level has been reported as a potential biomarker of lymph node metastasis and its expression has been linked to promoting migration and invasion of breast cancer cells. It has also been reported that correlations between decreased miRNA-373 expression and BC relapse.

However, findings often differed from each other due to different experiment design, study cohorts or disease status.

ELIGIBILITY:
Inclusion Criteria:

* Female age 20 years or older
* documented diagnosis of breast cancer based on physical examination, imaging and histopathology
* possibility of obtaining blood samples from the subject.

Exclusion Criteria:

* All patients with prior history of exposure to chemotherapy, radiotherapy or hormonal therapy .
* patients with other malignancies.
* patients with chronic inflammatory diseases.
* patients with missed documentation for histopathological diagnosis of breast cancer.

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This is a case control hospital-based study will conduct on women divided into two groups:
  Group A (patient group) : included patients with BC admitted to department of medical Oncology, South Egypt Cancer Institute, Assiut University. Whereas,
  Group B (control group) : included controls age-matched , sex-matched and apparently healthy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Assess serum miRNA-373 and miRNA-425-5p expression in patients with breast cancer. | baseline
  compare level of serum miRNA-373 and miRNA-425-5p expression in breast cancer patients with that of normal control in aim to help in diagnosis of BC patients and staging them

SECONDARY OUTCOMES:
Explore correlations of serum miRNA-373 and miRNA-425-5p expression in breast cancer patients with clinicopathological documented data including staging, grading and tumor receptors. | baseline
  aim to find significant correlations help in future diagnosis and treatment .

REFERENCES:
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Yalcin B. Staging, risk assessment and screening of breast cancer. Exp Oncol. 2013 Dec;35(4):238-45. PMID 24382431
- [Background] Autier P, Boniol M. Mammography screening: A major issue in medicine. Eur J Cancer. 2018 Feb;90:34-62. doi: 10.1016/j.ejca.2017.11.002. Epub 2017 Dec 20. PMID 29272783
- [Background] Matsen CB, Neumayer LA. Breast cancer: a review for the general surgeon. JAMA Surg. 2013 Oct;148(10):971-9. doi: 10.1001/jamasurg.2013.3393. PMID 23986370
- [Background] Aalami AH, Pouresmaeil V, Amirabadi A, Mojahed FH, Rad MQ, Sahebkar A. Evaluation of the Diagnostic Properties of Serum hsa-miR-223-5p in the Detection of Gastric Cancer: A Case-Control Study. Anticancer Agents Med Chem. 2020;20(7):800-808. doi: 10.2174/1871520620666200204100602. PMID 32013852
- [Background] Zhou Y, Sheng B, Xia Q, Guan X, Zhang Y. Association of long non-coding RNA H19 and microRNA-21 expression with the biological features and prognosis of non-small cell lung cancer. Cancer Gene Ther. 2017 Aug;24(8):317-324. doi: 10.1038/cgt.2017.20. Epub 2017 Aug 11. PMID 28799568
- [Background] Eichelser C, Flesch-Janys D, Chang-Claude J, Pantel K, Schwarzenbach H. Deregulated serum concentrations of circulating cell-free microRNAs miR-17, miR-34a, miR-155, and miR-373 in human breast cancer development and progression. Clin Chem. 2013 Oct;59(10):1489-96. doi: 10.1373/clinchem.2013.205161. Epub 2013 Jun 7. PMID 23748853
- [Background] Mangolini A, Ferracin M, Zanzi MV, Saccenti E, Ebnaof SO, Poma VV, Sanz JM, Passaro A, Pedriali M, Frassoldati A, Querzoli P, Sabbioni S, Carcoforo P, Hollingsworth A, Negrini M. Diagnostic and prognostic microRNAs in the serum of breast cancer patients measured by droplet digital PCR. Biomark Res. 2015 Jun 6;3:12. doi: 10.1186/s40364-015-0037-0. eCollection 2015. PMID 26120471
- [Background] Zhang LF, Zhang JG, Zhou H, Dai TT, Guo FB, Xu SY, Chen Y. MicroRNA-425-5p promotes breast cancer cell growth by inducing PI3K/AKT signaling. Kaohsiung J Med Sci. 2020 Apr;36(4):250-256. doi: 10.1002/kjm2.12148. Epub 2019 Nov 5. PMID 31688991
- [Background] Huang Q, Gumireddy K, Schrier M, le Sage C, Nagel R, Nair S, Egan DA, Li A, Huang G, Klein-Szanto AJ, Gimotty PA, Katsaros D, Coukos G, Zhang L, Pure E, Agami R. The microRNAs miR-373 and miR-520c promote tumour invasion and metastasis. Nat Cell Biol. 2008 Feb;10(2):202-10. doi: 10.1038/ncb1681. Epub 2008 Jan 13. PMID 18193036
- [Background] Inns J, James V. Circulating microRNAs for the prediction of metastasis in breast cancer patients diagnosed with early stage disease. Breast. 2015 Aug;24(4):364-9. doi: 10.1016/j.breast.2015.04.001. Epub 2015 May 6. PMID 25957467
- [Background] Pimentel F, Bonilla P, Ravishankar YG, Contag A, Gopal N, LaCour S, Lee T, Niemz A. Technology in MicroRNA Profiling: Circulating MicroRNAs as Noninvasive Cancer Biomarkers in Breast Cancer. J Lab Autom. 2015 Oct;20(5):574-88. doi: 10.1177/2211068214561788. Epub 2014 Dec 18. PMID 25524488
- [Background] Hosseini Mojahed F, Aalami AH, Pouresmaeil V, Amirabadi A, Qasemi Rad M, Sahebkar A. Clinical Evaluation of the Diagnostic Role of MicroRNA-155 in Breast Cancer. Int J Genomics. 2020 Sep 7;2020:9514831. doi: 10.1155/2020/9514831. eCollection 2020. PMID 32964011
- [Background] Swellam M, El Magdoub HM, Hassan NM, Hefny MM, Sobeih ME. Potential diagnostic role of circulating MiRNAs in breast cancer: Implications on clinicopathological characters. Clin Biochem. 2018 Jun;56:47-54. doi: 10.1016/j.clinbiochem.2018.04.013. Epub 2018 Apr 19. PMID 29679553
- See also: The Global Cancer Observatory — https://gco.iarc.fr/